CLINICAL TRIAL: NCT02977117
Title: The Effect of Increasing Dialysate Magnesium on Serum Calcification Propensity in Subjects With End-Stage Renal Disease Treated With Haemodialysis - A Randomised Clinical Trial
Brief Title: The Effect of Increasing Dialysate Magnesium on Calcification Propensity in Subjects on Haemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iain Bressendorff (Other)
Responsible Party: Sponsor-Investigator, Iain Bressendorff, MD, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Nordsjaellands Hospital
Record Dates: First submitted 2016-11-27; First posted 2016-11-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Endstage Renal Disease
Keywords: magnesium; ectopic calcification; chronic kidney disease - mineral and bone disorder; serum calcification propensity
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialysate magnesium 1.0 mmol/L (Experimental): Increase dialysate magnesium from 0.5 mmol/L to 1.0 mmol/L.
  Interventions: Other: Dialysate magnesium (1.0 mmol/L)
- Dialysate magnesium 0.5 mmol/L (Active Comparator): Maintain dialysate magnesium at 0.5 mmol/L.
  Interventions: Other: Dialysate magnesium (0.5 mmol/L)

INTERVENTIONS:
Other: Dialysate magnesium (1.0 mmol/L) — Dialysate magnesium will be increased from 0.5 mmol/L to 1.0 mmol/L for 4 weeks after which subjects will return to dialysate magnesium 0.5 mmol/L for 2 weeks observation.
  Arms: Dialysate magnesium 1.0 mmol/L
Other: Dialysate magnesium (0.5 mmol/L) — Dialysate magnesium will be maintained at 0.5 mmol/L for the duration of the trial.
  Arms: Dialysate magnesium 0.5 mmol/L

SUMMARY:
The purpose of this trial is to examine the effect of increasing dialyse magnesium on serum calcification propensity in subjects with end-stage renal disease treated with haemodialysis.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) have a 20-fold increased risk of cardiovascular mortality compared to the general population. Arterial stiffness, likely due to vascular calcification (VC), has been shown to predict cardiovascular mortality in ESRD. Serum calcification propensity (T50) is a novel biomarker, which is believed to reflect the propensity toward ectopic calcification (e.g. VC). Increasing serum magnesium (sMg) should increase T50, which might in turn reduce the formation of VC in patients with ESRD. A cheap and easy way of achieving this would be to increase the concentration of Mg in the dialysate (dMg) of patients with ESRD treated with haemodialysis (HD).

The investigators wish to conduct a randomised controlled double-blind clinical trial to examine whether increasing dMg will improve T50 in subjects with ESRD treated with HD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Treatment with maintenance haemodialysis for more than 3 months.
* Dialysate magnesium of 0.5 mmol/L (standard concentration).
* Serum magnesium < 1.2 mmol/L on average of previous measurements within the last 3 months.
* Women of childbearing age must be actively using contraceptive therapy (p-pills, estrogen depots or intrauterine device) as well as have a negative pregnancy test.
* Written informed consent.

Exclusion Criteria:

* Treatment with peritoneal dialysis.
* Parathyroid hormone > 66 ρmol/L.
* Previous parathyroidectomy.
* Current treatment with magnesium containing medication or supplements.
* Other diseases or conditions, which, in the opinion of the site investigator, would prevent participation in or completion of the trial.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Between-group difference in serum calcification propensity at follow-up | 4 weeks

SECONDARY OUTCOMES:
Within-group change in serum calcification propensity | 2 weeks
Within-group change and between-group difference in serum magnesium | 4 weeks
Change in serum magnesium after intervention | 2 weeks
Within-group change and between-group difference in serum parathyroid hormone | 4 weeks
Change in serum parathyroid hormone after intervention | 2 weeks
Change in fibroblast growth factor 23 during intervention | 4 weeks
Incidence of intradialytic hypotension during intervention | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Iain Bressendorff, Hillerød, Denmark